CLINICAL TRIAL: NCT00558662
Title: Randomized Controlled Clinical Study to Assess the Clinical Efficacy of the 3M™ Coban™ 2 Layer Compression System Compared to a Short-stretch Compression Bandage in the Treatment of Venous Leg Ulcers
Brief Title: Randomized Clinical Trial (RCT) to Compare the Efficacy of Coban 2 Versus SSB in the Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EU Study No-05-000003
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Venous Ulcer
Keywords: compression therapy; venous leg ulcer; sub bandage pressure
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Coban 2 Layer Compression System
  Interventions: Device: Coban 2
- 2 (Active Comparator): Short-Stretch Bandage
  Interventions: Device: SSB

INTERVENTIONS:
Device: Coban 2 — Bandages will be changed after a wear time of seven days, or in case of product or non-product related reason, which would require a dressing or bandage change.
  Other Names: Coban 2 Layer Compression System
  Arms: 1
Device: SSB — Bandages will be changed after a wear time of seven days, or in case of product or non-product related reason, which would require a dressing or bandage change.
  Other Names: Rosidal K; Rosidal soft
  Arms: 2

SUMMARY:
The study purpose is to compare healing rates, cost effectiveness, quality of life and safety of 12 week compression therapy for the treatment of venous leg ulcers with the 3M™ Coban™ 2 Layer Compression System versus short-stretch compression bandage.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 18 years or older
* Subjects having a venous leg ulcer (stage C6 according CEAP classification, venous pathology proved by the presence of reflux (Pr)), which is at least 1 cm in any dimension but not larger than 10 cm in any dimension and has at least 5 cm distance to additional ulcers.
* Subjects who are co-operative, willing to give written informed consent prior to study entry, and willing to comply with the study protocol.
* Subjects who are able to understand and answer questionnaire items.
* Subjects who can walk (with or without a walking aid).
* Subjects who have an ABPI (ankle brachial pressure index) of treated leg greater or equal to 0,8 as measured within four weeks prior to enrollment.
* Subjects with venous incompetence as defined by reflux longer than 1,0 second in at least one of the following sites: groin [femoral vein, junction of GSV], mid thigh medial [GSV], hollow of the knee [popliteal vein, junction of SSV], mid calf [SSV] in the standing position, measured by Doppler, preferably by duplex within the last 12 month without following active treatment of venous reflux.

Exclusion Criteria:

* Subjects with an ABPI < 0.8 as measured within four weeks prior to enrollment.
* Subjects whose condition, in the opinion of the investigator, does not require or allow for compression therapy.
* Subjects where the potential study ulcer is infected, i.e. showing signs of clinical infection (not contamination) as evidenced by purulent, malodorous, or recent increase in drainage and/or peri-wound erythema or elevated temperature.
* Subjects receiving any systemic antibiotics.
* Subjects with diagnosed cancerous ulceration.
* Subjects with diabetic foot ulcers (do not exclude diabetics).
* Subjects with circumferential wounds.
* Subjects who started or significantly changed treatment with mood altering substances (e.g. antidepressant drugs) within two weeks prior to enrollment.
* Subjects who are participating in any prospective clinical study that can potentially interfere with this study.
* Subjects who are, in the opinion of the clinical investigator, unsuitable for enrollment in this study, for reasons not specified in the exclusion criteria.
* Subjects with known allergies against the following products: Coban 2 Layer Compression System, Rosidal K, Rosidal soft, Tegaderm Foam, Cavilon NSBF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
- venous leg ulcer healing | 12 weeks

SECONDARY OUTCOMES:
- wound size reduction - HRQoL - treatment-cost based on material consumption and visit costs - sub-bandage pressure measurements - AE/SAE | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Vanscheidt, Prof MD PhD, Study Chair; Eberhard Rabe, Prof. MD PhD, Principal Investigator — Klnik und Poliklinik für Dermatologie der Universität Bonn; Joachim Dissemond, MD PhD, Principal Investigator — Universitätsklinik Essen; Markus Stücker, MD PhD, Principal Investigator — Klinik für Dermatologie der Rhur Universität Bochum; Keith Harding, MB, MRCGP, FRCS, Principal Investigator — Wound Healing Research Unit; Jost van der Kleij, MD, PhD, Principal Investigator — Atrium Medisch Centrum Parkstad in Heerlen; Karl-Heinz Konz, MD PhD, Principal Investigator — Kliniken Maria Hilf Mönchengladbach; Jose Schroijen, MD PhD, Principal Investigator — Department of Dermatology, Ziekenhuis de Lievensberg; Dinanda Kolbach, MD PhD, Principal Investigator — Dr. Kolbach Kliniek; Karin Timm, Principal Investigator — IJsselland Hospital; Gill Wicks, Principal Investigator — Tissue Viability; Sylvie Hampton, MA BSc (Hons) DpSN RGN, Principal Investigator — Tissue Viability; Helger Stege, MD PhD, Principal Investigator — Klinikum Lippe-Lemgo; Rik Couvreur, MD, PhD, Principal Investigator — Military Hospital Queen Astrid; Toon Sabbe, MD, PhD, Principal Investigator — AZ alma Eeklo; Rudi Vossaert, MD, PhD, Principal Investigator — Wound Centre AZ St. Elisabeth
Locations (16):
- Belgium (3):
  - Wound Centre AZ St. Elisabeth, Zottegem, Godveerdegemstraat 69
  - AZ Alma Eeklo, Eeklo, Moeie 13
  - Military Hospital Queen Astrid, Brussels, Neder-Over-Heembeek
- Germany (6):
  - Klinik für Dermatologie der Rhr Universität Bochum - Venenzentrum der dermatologischen und gefäßchirurgischen Kliniken, Bochum
  - Klinik und Poliklinik für Dermatologie der Universität Bonn, Bonn
  - Universitätsklinikum Essen, Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Essen
  - Prof. Vanscheidt, MD, PhD, Freiburg im Breisgau
  - Klinikum Lippe_lemgo, Lemgo
  - Kliniken Maria Hilf, Mönchengladbach
- Netherlands (4):
  - Ziekenhuis de Lievensberg, Department of Dermatology, Bergen op Zoom
  - IJsselland Hospital, Capelle aan den IJssel
  - Atrium Medisch Centrum Parkstad in Heerlen, Heerlen
  - Dr. Kolbach Kliniek, Maastricht
- United Kingdom (3):
  - Wound Healing Research unit, Cardiff Medicentre, Cardiff
  - Tissue Viability, Eastbourne
  - Trowbridge Community Hospital, Trowbridge